CLINICAL TRIAL: NCT04807101
Title: A Randomized Study of Midazolam and Fentanyl Versus Midazolam Alone for Sedation in Gastrointestinal Endoscopy
Brief Title: Sedation Regimens in GI Endoscopy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Greg S Cohen MD LLC (Other)
Responsible Party: Principal Investigator, Greg Cohen, Clinical Associate Professor of Medicine, Greg S Cohen MD LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU#: 00214212
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia; Endoscopy; Colonoscopy; Conscious Sedation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- midazolam and fentanyl (No Intervention): Patients in this arm will receive standard conscious sedation with midazolam and fentanyl
- midazolam alone (Experimental): Patients in this arm will receive conscious sedation with medazepam alone
  Interventions: Drug: midazolam alone

INTERVENTIONS:
Drug: midazolam alone — elimination of fentanyl from conscious sedation
  Arms: midazolam alone

SUMMARY:
This is a noninferiority study designed to examine whether conscious sedation with midazolam alone results in efficacy and safety that is not inferior to the combination of midazolam and fentanyl. English-speaking patients ≥18 years old and ≤75 years old presenting for GI endoscopy planned with conscious sedation using midazolam and fentanyl, will be randomized 1:1 to single agent sedation with midazolam or combination sedation with midazolam and fentanyl. Participants will be blinded to the choice of sedation. Sedation quality and adverse events will be measured with a validated patient-centered measure of procedural sedation quality, the PROcedural Sedation Assessment Survey (PROSAS) [Leffler, et al. Gastrointest Endosc. 2015;81(1):194-203]. Endoscopic quality measures in the 2 study groups will be collected by retrospective chart review, as an additional metric to ensure the quality of the procedure is not compromised by the choice of sedation.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* Patients ≥18 years old and ≤75 years old
* Outpatients presenting for EGD and/or colonoscopy planned with conscious sedation using midazolam and fentanyl
* Patients presenting for endoscopic procedures with no GI fellow or trainee involvement in the procedure

Exclusion Criteria:

* Patients with an allergy or prior adverse event to either fentanyl or midazolam
* Patients who have previously not tolerated endoscopy with conscious sedation and require monitored anesthesia care (MAC)
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Vulnerable populations, including cognitively impaired adults and adults who are otherwise unable to consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Started | 152 | 148
Completed | 152 | 148
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam and Fentanyl | Midazolam Alone | Total
Number analyzed (Participants) | 152 | 148 | 300
Age, Continuous [Median (Standard Deviation); unit: years] | 52.3 (11.1) | 52.3 (10.4) | 52.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 61 | 133
  Male | 80 | 87 | 167
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 152 | 148 | 300

OUTCOME MEASURES:

1. Primary Outcome: Pain Felt During the Procedure
Description: Level of discomfort during the procedure as assessed by the previously validated PROcedural Sedation Assessment Survey (PROSAS) questionnaire [Leffler, et al. Gastrointest Endosc. 2015;81(1):194-203]. The patient will answer the question "How much discomfort did you experience during the procedure?" A visual analog scale will be used ranging from 0 to 10 with higher numbers indicating more pain.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
score on a scale | 0.29 (1.2) | 0.30 (1.1)

2. Primary Outcome: Adequacy of Sedation
Description: Adequacy of sedation as assessed by the previously validated PROcedural Sedation Assessment Survey (PROSAS) questionnaire [Leffler, et al. Gastrointest Endosc. 2015;81(1):194-203]. The patient will answer the question "If having this procedure again in the future, how much sedation would you prefer to have?" A visual analog scale will be used ranging from -5 to 5, with lower numbers indicating a preference for less sedation in the future and higher numbers indicating a preference for more sedation in the future.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
score on a scale | -0.28 (0.94) | -0.094 (0.78)

3. Secondary Outcome: Patient Reported Nausea
Description: Patient reported nausea as assessed by a yes or no answer to the question "Do you have any nausea now?"
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
Participants | 1 | 1

4. Secondary Outcome: Adverse Events
Description: Oxygen desaturation, hypotension, or any other event requiring the procedure to be interrupted
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
Participants | 1 | 2

5. Secondary Outcome: Cecal Intubation Rate
Description: cecal intubation rate for the 2 arms of the study will be assessed by retrospective chart review
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
Participants | 152 | 148

6. Secondary Outcome: Cecal Intubation Time
Description: time to reach the cecum for the 2 arms of the study will be assessed by retrospective chart review
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
minutes | 6.97 (3.10) | 7.99 (3.66)

7. Secondary Outcome: Colonoscopy Withdrawal Time
Description: Colonoscopy withdrawal time for the 2 arms of the study will be assessed by retrospective chart review
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
minutes | 16.44 (4.01) | 16.29 (4.34)

8. Secondary Outcome: Adenoma Detection Rate
Description: Adenoma detection rate for the 2 arms of the study will be assessed by retrospective chart review
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
Number analyzed (Participants) | 152 | 148
Participants | 58 | 54

ADVERSE EVENTS:
Time Frame: 1 day
Description: oxygen desaturation, hypotension, or any other event requiring the procedure to be interrupted
Arm/Group | Midazolam and Fentanyl | Midazolam Alone
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/148
Other Adverse Events (participants affected / at risk) | 1/152 | 2/148
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam and Fentanyl (N=152) | Midazolam Alone (N=148)
procedure interrupted due to pain (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT04807101/Prot_SAP_000.pdf